CLINICAL TRIAL: NCT06398977
Title: Dapagliflozin Delays the Loss of Residual Renal Function in Patients Undergoing Peritoneal Dialysis: A Single-Center Randomized Open-Label Study
Brief Title: Dapagliflozin Delays the Loss of Renal Function in Peritoneal Dialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jin Chen, vice professor, Sichuan Academy of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DDLR-PD
Record Dates: First submitted 2024-04-16; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Dialysis Complication; Renal Function Aggravated; Sodium-glucose Co-transporter-2 Inhibitors
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dagliflozin group (Active Comparator): Patients in this group were treated with dagliflozin 10 mg, oral once daily, for 24 weeks, in addition to receiving basic treatments such as peritoneal dialysis and antihypertensive and hypoglycemic therapy.
  Interventions: Drug: Dapagliflozin
- Control group (No Intervention): This group of patients received peritoneal dialysis and basic treatments such as antihypertensive and hypoglycemic therapy.

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin10MG, PO once daily
  Other Names: dagliflozin
  Arms: Dagliflozin group

SUMMARY:
This study aims to explore the role of dagliflozin in preserving the residual renal function(RRF) in peritoneal dialysis (PD) patients.

DETAILED DESCRIPTION:
Residual renal function (RRF) plays the role of removing water and body metabolic wastes, as well as secretion of erythropoietin and promotion of vitamin D absorption, which can maintain the stability of the internal environment. Several studies have demonstrated that preservation of RRF in PD patients reduces complications, increases dialysis adequacy and decreases mortality. In addition, residual renal function is an important factor in the technique survival. Methods to protect residual renal function in peritoneal dialysis patients include controlling blood pressure, controlling blood glucose, adjusting dialysis prescription, and using renin-angiotensin inhibitors. However, the above methods currently play only a limited role.

Sodium-dependent glucose transporters 2 (SGLT2) inhibitors are drugs used in the treatment of type 2 diabetes mellitus that inhibit the reabsorption of glucose by the kidneys, causing glucose to be excreted in the urine and lowering blood glucose. Studies have demonstrated that SGLT2 inhibitors also attenuate renal tubular injury, reduce the excretion of proteinuria, and have a protective effect on RRF in non-dialysis patients with chronic kidney disease. However, there are no clinical studies demonstrating whether the use of SGLT2 inhibitors in peritoneal dialysis patients is renal protective.

In light of this, this study introduces dagliflozin orally to PD patients over a 24-week period to explore its protective effects on RRF and cardiac health, with participants being randomly divided into a dagliflozin group and a control group. The results of this study will be beneficial in informing the clinical practice of SGLT2 inhibitors and improving dialysis outcomes in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD duration between 1 month and 3 months.
* Patients aged between 18 and 75 years.
* Voluntary signing of informed consent.
* Stable use of a maximum tolerated dose of RAAS inhibitors for one month if hypertension is present.
* Daily urine output ≥ 400ml/day.
* Stable PD prescription for one month.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with type 1 diabetes mellitus.
* Patients with type 2 diabetes mellitus who have experienced diabetic ketoacidosis in the past.
* Patients with chronic liver disease, including non-alcoholic fatty liver disease, cirrhosis, ALT > 120 IU/L, and other clinically confirmed severe liver diseases.
* Patients with more than 2 episodes of urinary tract infection in the past six months.
* Patients with severe allergic reactions (rash or angioedema) to Dapagliflozin.
* Patients using the following medications: rifampicin, phenytoin.
* Patients with malignant tumors.
* Patients who developed peritonitis within one month.
* Patients undergoing combined hemodialysis treatment.
* Patients with a willingness for kidney transplantation within six months.
* Patients with a history of pancreatitis or pancreatic transplantation.
* Patients who experienced acute coronary syndrome or cerebrovascular events within one month.
* Hemoglobin level less than 90g/L.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 24 urine volume | Baseline, 2,12 and 24 weeks.
  The total amount of urine excreted over a 24-hour period. The patient's urine output was measured continuously for 2 days, and the average volume was calculated, with the unit being millilitres.

SECONDARY OUTCOMES:
Change in renal Kt/Vurea | Baseline, 2, 12 and 24 weeks.
  A measure used in peritoneal dialysis therapy to assess adequacy, representing the renal clearance of urea (K) over time (t) normalized to body water volume (V).
Change in BNP（Brain natriuretic peptide） | Baseline, 2, 12 and 24 weeks.
  Concentration of serum BNP which could assess cardiac function.
Change in EF% | Baseline and 24 weeks.
  The ejection fraction (EF%) value was measured using echocardiography by the hospital's ultrasound department, with all ultrasound examinations conducted by two attending physicians.
Change in ultrafiltration | Baseline, 2, 12 and 24 weeks.
  The total amount of water removed from the body through dialysis each day.
Change in HbA1C （Hemoglobin A1C) rate | Baseline, 12 and 24 weeks.
  Rate of Glycated Hemoglobin (HbA1C) as an Indicator of Long-term Glycemic Control in Serum.
Change in serum sodium concentration | Baseline, 2, 12 and 24 weeks.
  Concentration of sodium ions in the blood.
Change in urinary sodium concentration | Baseline, 2, 12 and 24 weeks.
  The concentration of sodium in the 24-hour urine.
Change in dialysate sodium concentration | Baseline, 2, 12 and 24 weeks.
  The concentration of sodium in the 24-hour dialysate.
Change in urinary glucose concentration | Baseline, 2, 12 and 24 weeks.
  The concentration of glucose in the 24-hour urine.
Change in blood pressure | Baseline, 2, 12 and 24 weeks.
  The bloody pressure of the patient in the morning.
Change in body weight | Baseline, 2, 12 and 24 weeks.
  The weight of the patient is measured on an empty stomach without containing dialysate.
Episodes of peritonitis | 24 weeks.
  The number of episodes of a patient during the trial.
Hospitalization | 24 weeks.
  The number of patients admitted to hospital during the trial.
Time of dropout PD | 24 weeks.
  The point in time at which a patient either discontinues PD treatment or experiences death during the trail.
Concentration in Dapagliflozin 3-O-Glucuronide in urine | Baseline, 2, 12 and 24 weeks.
  Concentration of Dapagliflozin 3-O-Glucuronide in urine indicating Dapagliflozin metabolic activity.
Concentration in Dapagliflozin 3-O-Glucuronide in dialysate | Baseline, 2, 12 and 24 weeks.
  Concentration of Dapagliflozin 3-O-Glucuronide in dialysate reflecting Dapagliflozin metabolism.
concentration of Dapagliflozin 3-O-Glucuronide in serum | Baseline, 2, 12 and 24 weeks.
  Concentration of Dapagliflozin 3-O-Glucuronide in serum reflecting Dapagliflozin metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Chen, MD, Principal Investigator — Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospita, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Wal WM, Noordzij M, Dekker FW, Boeschoten EW, Krediet RT, Korevaar JC, Geskus RB; Netherlands Cooperative Study on the Adequacy of Dialysis Study Group (NECOSAD). Full loss of residual renal function causes higher mortality in dialysis patients; findings from a marginal structural model. Nephrol Dial Transplant. 2011 Sep;26(9):2978-83. doi: 10.1093/ndt/gfq856. Epub 2011 Feb 11. PMID 21317411
- [Background] Bargman JM, Thorpe KE, Churchill DN. Relative contribution of residual renal function and peritoneal clearance to adequacy of dialysis: a reanalysis of the CANUSA study. J Am Soc Nephrol. 2001 Oct;12(10):2158-2162. doi: 10.1681/ASN.V12102158. PMID 11562415
- [Background] Bello AK, Okpechi IG, Osman MA, Cho Y, Cullis B, Htay H, Jha V, Makusidi MA, McCulloch M, Shah N, Wainstein M, Johnson DW. Epidemiology of peritoneal dialysis outcomes. Nat Rev Nephrol. 2022 Dec;18(12):779-793. doi: 10.1038/s41581-022-00623-7. Epub 2022 Sep 16. PMID 36114414
- [Background] Parving H-H, Lambers-Heerspink H, de Zeeuw D. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Nov 3;375(18):1800-1. doi: 10.1056/NEJMc1611290. No abstract available. PMID 28106974
- [Background] Persson F, Rossing P, Vart P, Chertow GM, Hou FF, Jongs N, McMurray JJV, Correa-Rotter R, Bajaj HS, Stefansson BV, Toto RD, Langkilde AM, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Efficacy and Safety of Dapagliflozin by Baseline Glycemic Status: A Prespecified Analysis From the DAPA-CKD Trial. Diabetes Care. 2021 Aug;44(8):1894-1897. doi: 10.2337/dc21-0300. Epub 2021 Jun 28. PMID 34183431
- [Background] Zelniker TA, Wiviott SD, Raz I, Im K, Goodrich EL, Furtado RHM, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Sabatine MS. Comparison of the Effects of Glucagon-Like Peptide Receptor Agonists and Sodium-Glucose Cotransporter 2 Inhibitors for Prevention of Major Adverse Cardiovascular and Renal Outcomes in Type 2 Diabetes Mellitus. Circulation. 2019 Apr 23;139(17):2022-2031. doi: 10.1161/CIRCULATIONAHA.118.038868. PMID 30786725
- [Background] Birkeland KI, Jorgensen ME, Carstensen B, Persson F, Gulseth HL, Thuresson M, Fenici P, Nathanson D, Nystrom T, Eriksson JW, Bodegard J, Norhammar A. Cardiovascular mortality and morbidity in patients with type 2 diabetes following initiation of sodium-glucose co-transporter-2 inhibitors versus other glucose-lowering drugs (CVD-REAL Nordic): a multinational observational analysis. Lancet Diabetes Endocrinol. 2017 Sep;5(9):709-717. doi: 10.1016/S2213-8587(17)30258-9. Epub 2017 Aug 3. PMID 28781064
- [Background] Persson F, Nystrom T, Jorgensen ME, Carstensen B, Gulseth HL, Thuresson M, Fenici P, Nathanson D, Eriksson JW, Norhammar A, Bodegard J, Birkeland KI. Dapagliflozin is associated with lower risk of cardiovascular events and all-cause mortality in people with type 2 diabetes (CVD-REAL Nordic) when compared with dipeptidyl peptidase-4 inhibitor therapy: A multinational observational study. Diabetes Obes Metab. 2018 Feb;20(2):344-351. doi: 10.1111/dom.13077. Epub 2017 Sep 8. PMID 28771923
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] Lui SL, Yung S, Yim A, Wong KM, Tong KL, Wong KS, Li CS, Au TC, Lo WK, Ho YW, Ng F, Tang C, Chan TM. A combination of biocompatible peritoneal dialysis solutions and residual renal function, peritoneal transport, and inflammation markers: a randomized clinical trial. Am J Kidney Dis. 2012 Dec;60(6):966-75. doi: 10.1053/j.ajkd.2012.05.018. Epub 2012 Jul 25. PMID 22835900
- [Result] Li T, Wilcox CS, Lipkowitz MS, Gordon-Cappitelli J, Dragoi S. Rationale and Strategies for Preserving Residual Kidney Function in Dialysis Patients. Am J Nephrol. 2019;50(6):411-421. doi: 10.1159/000503805. Epub 2019 Oct 18. PMID 31630148
- [Result] Mosenzon O, Wiviott SD, Cahn A, Rozenberg A, Yanuv I, Goodrich EL, Murphy SA, Heerspink HJL, Zelniker TA, Dwyer JP, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Kato ET, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS, Raz I. Effects of dapagliflozin on development and progression of kidney disease in patients with type 2 diabetes: an analysis from the DECLARE-TIMI 58 randomised trial. Lancet Diabetes Endocrinol. 2019 Aug;7(8):606-617. doi: 10.1016/S2213-8587(19)30180-9. Epub 2019 Jun 10. PMID 31196815
- [Result] Barreto J, Borges C, Rodrigues TB, Jesus DC, Campos-Staffico AM, Nadruz W, Luiz da Costa J, Bueno de Oliveira R, Sposito AC. Pharmacokinetic Properties of Dapagliflozin in Hemodialysis and Peritoneal Dialysis Patients. Clin J Am Soc Nephrol. 2023 Aug 1;18(8):1051-1058. doi: 10.2215/CJN.0000000000000196. Epub 2023 May 25. PMID 37227937

DOCUMENTS (1):
  • Informed Consent Form (2024-02-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT06398977/ICF_000.pdf